CLINICAL TRIAL: NCT02424552
Title: EVITA Trial: Effect of VItamin D as add-on Therapy for Vitamin D Insufficient Patients With Severe Asthma: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effect of Vitamin D as add-on Therapy for Vitamin D Insufficient Patients With Severe Asthma
Acronym: EVITA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: recruitment problems
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, PD Dr. Stephanie Korn, Principal Investigator, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-003; 2014-002363-15 (EudraCT Number)
Record Dates: First submitted 2015-04-14; First posted 2015-04-23 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Asthma
Keywords: severe asthma; vitamin D; treatment
MeSH Terms: conditions — Asthma | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Experimental): Initial single dose 100000 IU, beginning from the second day 4000 IU/day for 24 weeks
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): Amount of Placebo capsules corresponding to initial single dose of Vitamin D3, beginning from the second day amount of capsules corresponding to daily dose of Vitamin D for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Initial single dose 100000 IU, beginning from the second day 4000 IU/day for 24 weeks.
  Other Names: Cholecalciferol
  Arms: Vitamin D3
Drug: Placebo — Filling material: lactose monohydrate, cellulose, magnesium stearate
  Arms: Placebo

SUMMARY:
The purpose of the EVITA trial is to compare the effects of vitamin D therapy with placebo on reducing the dose of inhaled or oral corticosteroids in patients with severe asthma and vitamin D insufficiency.

DETAILED DESCRIPTION:
Patients with severe asthma represent the greatest unmet medical need among the asthmatic population, in particular due to their high risk of severe exacerbations. A substantial proportion of these patients does not achieve asthma control despite even high-dose ICS and LABA treatment, necessitating add-on therapy. For these patients oral corticosteroids (OCS) are a preferred treatment modality, which will inevitably lead to severe side effects. A high Proportion of patients with severe Asthma are Vitamin D insufficient (< 30 ng/ml). It is therefore tempting to speculate that vitamin D substitution in vitamin D insufficient patients who continue to experience suboptimal asthma control on ICS and LABA or ICS/LABA plus OCS treatment may boost corticosteroid responsiveness, thereby potentially reducing corticosteroid dose requirements and improving key parameters of asthma control.

The present study is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of treatment with vitamin D at a dose of 4000 IU/day administered daily following a single loading dose of 100 000 IU upon study entry over a period of 24 weeks in patients with severe asthma and vitamin D insufficiency. During the study, all patients will remain on their existing maintenance asthma therapy throughout the study, in addition to the study treatment, while reducing inhaled or oral steroids according to study protocol. The study consists of a 2-week run-in period, a 24 week double-blind treatment period including a 12 week steroid stable phase and two steroid reduction phases, followed by a follow-up visit 4 weeks after last study medication intake. The active treatment arm in this study will be standard of care plus vitamin D (loading dose of 100 000 IU upon study entry, to be followed by 4000 IU/day for the rest of the study period) while the comparator arm will be standard of care plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age ≥ 18 years
* A pulmonary specialist documented diagnosis of severe asthma according to the Global Initiative for Asthma and the German Asthma Network (GAN, www.german-asthma-net.de)
* Treatment with long-acting β2-agonists (LABA) and inhaled corticosteroids (ICS) at a dose of at least 1000 µg beclomethasone (or equivalent) per day, - chronic oral corticosteroid (OCS) use is allowed Stable asthma medication for ≥1 month prior to screening (≥4 months for omalizumab)
* Asthma Control Questionnaire (ACQ-5) score ≥ 1.5
* Vitamin D insufficiency as defined by a serum vitamin D concentration of < 30 ng/ml but ≥ 10 ng/ml at screening

Exclusion Criteria:

* Patients on vitamin D substitution
* Current smokers or ex-smokers with a smoking history of more than 10 pack-years
* Pregnant or nursing women or women who intend to become pregnant during the study
* Known impaired renal function (GFR < 30 ml/min) and history of physician-diagnosed nephrolithiasis
* Use of other investigational drugs during the study or within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-03-09 (Actual)

PRIMARY OUTCOMES:
relative dose reduction of ICS or OCS at week 24 as assessed by total ICS or OCS dose | 24 weeks

SECONDARY OUTCOMES:
Exacerbations (rate of and time to first and subsequent exacerbations) as assessed by numbers of exacerbations | 24 weeks and 30 weeks
Asthma Control as assessed by ACQ score | at weeks 4, 8, 12, 14, 18, 20, 24, and 28
Asthma Quality of Life as assessed by the Mini-AQLQ score | at weeks 12, 18, 24 and 28
Pulmonary function test results as assessed by FEV1, FVC, IC, RV, TLC, and airway resistance | at weeks 4, 8, 12, 14, 18, 20, 24, and 28
Levels of vitamin D as assessed by serum concentrations | at weeks 12, 18, 24 and 28
Proportion of patients that achieved vitamin D sufficiency | at week 24
Assessment of safety and tolerability as assessed by number of adverse events | up to 30 weeks
Dyspnea as assessed by Baseline and Transition Dyspnea Indexes | at weeks 12, 18, 24 and 28

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Korn, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (9):
- Germany (9):
  - Pneumologische Gemeinschaftspraxis Dr. Rolke & Dr. Rückert, Aschaffenburg
  - Medizinische Klinik III für Pneumologie, allergologie, Schlaf- und Beatmungsmedizin, Berufsgenossenschaftliches Universitätsklinikum Bochum-Bergmannsheil GmbH, Bochum
  - IKF Pneumologie GmbH & Co.KG, Frankfurt
  - Pneumologisches Forschungsinstitut der LungenClinic Grosshansdorf, Großhansdorf
  - Studienzentrum KPPK GmbH, Koblenz
  - KLB - Gesundheitsforschung Lübeck GmbH, Lübeck
  - Pneumologie, III. Medizinische Klinik, Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Regensburg, Klinik und Poliklinik für Innere Medizin II/Pneumologie, Regensburg
  - Lungenpraxis Schleswig, Schleswig

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Korn S, Hubner M, Jung M, Blettner M, Buhl R. Severe and uncontrolled adult asthma is associated with vitamin D insufficiency and deficiency. Respir Res. 2013 Feb 22;14(1):25. doi: 10.1186/1465-9921-14-25. PMID 23432854
- [Background] Martineau AR, MacLaughlin BD, Hooper RL, Barnes NC, Jolliffe DA, Greiller CL, Kilpin K, McLaughlin D, Fletcher G, Mein CA, Hoti M, Walton R, Grigg J, Timms PM, Rajakulasingam RK, Bhowmik A, Rowe M, Venton TR, Choudhury AB, Simcock DE, Sadique Z, Monteiro WR, Corrigan CJ, Hawrylowicz CM, Griffiths CJ. Double-blind randomised placebo-controlled trial of bolus-dose vitamin D3 supplementation in adults with asthma (ViDiAs). Thorax. 2015 May;70(5):451-7. doi: 10.1136/thoraxjnl-2014-206449. Epub 2015 Feb 27. PMID 25724847
- [Background] Castro M, King TS, Kunselman SJ, Cabana MD, Denlinger L, Holguin F, Kazani SD, Moore WC, Moy J, Sorkness CA, Avila P, Bacharier LB, Bleecker E, Boushey HA, Chmiel J, Fitzpatrick AM, Gentile D, Hundal M, Israel E, Kraft M, Krishnan JA, LaForce C, Lazarus SC, Lemanske R, Lugogo N, Martin RJ, Mauger DT, Naureckas E, Peters SP, Phipatanakul W, Que LG, Sheshadri A, Smith L, Solway J, Sullivan-Vedder L, Sumino K, Wechsler ME, Wenzel S, White SR, Sutherland ER; National Heart, Lung, and Blood Institute's AsthmaNet. Effect of vitamin D3 on asthma treatment failures in adults with symptomatic asthma and lower vitamin D levels: the VIDA randomized clinical trial. JAMA. 2014 May;311(20):2083-91. doi: 10.1001/jama.2014.5052. PMID 24838406